CLINICAL TRIAL: NCT01553045
Title: Observational Study of the Variation in Health-related Quality of Life and Symptom Burden in Patients Accepted for Catheter Ablation of Atrial Fibrillation in Relation to Biomarkers, Intracardiac Pressures and Echocardiography.
Brief Title: Reasons for Variations in Health Related Quality of Life and Symptom Burden in Patients With Atrial Fibrillation
Acronym: SMURF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Hakan Walfridsson, Associate professor, M.D., University Hospital, Linkoeping
Other Study IDs: SMURF
Record Dates: First submitted 2012-02-02; First posted 2012-03-13 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Arrhythmias, Cardiac; Heart Failure, Systolic; Atrial Fibrillation
Keywords: symptom burden; atrial fibrillation; biomarkers; intracardiac pressures
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure, Systolic; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn from femoral vein, CS and LA (baseline sampling).
  Concerning sub-study: After the induction of AF and after the patient has maintained AF in 30 minutes blood samples will be drawn in the exact same way as before the induction in the intervention group.
  Patients who are going to be randomized to control group after the baseline blood sampling, are going to be monitored in about 30 minutes to examine whether they maintain sinus rhythm (SR) under that time. No intervention, clinical or experimental is going to be made during that time. After those 30 minutes, blood samples are going to be drawn in the exact same way as before.
  Blood to be analyzed for biomarkers will be froozen to -70 degress and analyzed when the study is completed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- atrial fibrillation, catheter ablation: Patients referred for ablation of atrial fibrillation

SUMMARY:
Atrial fibrillation is the most common cardiac arrhythmia. There is a large variation in symptoms; from almost none to severe but the reason for this is unclear.

The investigators aim to find correlations between symptom burden and intracardiac pressure, biomarkers and findings with echocardiography in order to find alternative means of treatment.

It is even intended to study the neurohormonal activation directly after the atrial fibrillation (AF) initiation in patients eligible for AF radiofrequency ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and more than 1 % of the population suffers from AF, it is an independent risk factor for ischemic stroke One major unresolved issue concerning AF is the large variety in symptoms. In some AF is diagnosed accidentally while in others symptoms are severe and disabling.

It is known that B-type natriuretic peptide (BNP) and atrial natriuretic peptide (ANP) is stored in nodules in the atrial and ventricular myocytes and is produced in response to increased 'afterload' and 'preload' to restore and maintain cardiovascular homeostasis. Vasopressin (AVP), a non-cardiac plasma marker of cardiovascular disease, is released from the neurohypophysis in response to changes in plasma osmolality and is involved in osmoregulation and cardiovascular homeostasis. Adrenomodullin originates primarily in endothelial cells where cellular stress, ischaemia and hypoxia result in an increased production.

It is well-known that the concentrations of the natriuretic peptides are elevated in patients with AF and that the plasma concentrations decreased after conversion to sinus rhythm (SR). Yet their reaction when AF initiates is totally unknown. Moreover the role of ADM and AVP-hormonal system has not been researched in this category of patients.

Patients scheduled for catheter ablation of AF for the first time will be included; all with symptoms varying from moderate to severe. Using four health related quality of life forms the impact of AF on symptoms will be evaluated. Patients will be investigated with echocardiography, invasive hemodynamics and measurement of the levels of peptide indicators of heart failure and/or impact on myocardial function. Patients will also be categorized according to metabolic profile.

The information on this subject is scarce. Hemodynamic data is old and not correlated to symptoms. Effective and validated means of measuring health related quality of life including symptoms burden are relatively new tools. The aim is to find correlations between the impact on health related quality of life and parameters from echocardiographic measurements, from analysis of biomarkers (peptides) and from analysis of the metabolic profile.

In order to study the response of these four different neurohormonal systems (represented by NT-proBNP, MR-proANP, MR-proADM, copeptin) after the initiation of AF, a randomized interventional clinical sub-study is to be performed where the eligible population of SMURF main study can be randomized to AF induction or to control if freedom from AF is confirmed with thumb-ecg during the last 4 days before ablation. 45 patients are to be included to the sub-study with 2:1 allocation ratio with simple randomization.

If such correlations can be found alternate means for symptoms relief in AF patients can be identified and further ahead implemented in general health care.

The sub-study can give us a better insight on the AF initiation and the activation of different neurohormonal systems, an areas which is not well investigated.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or paroxysmal atrial fibrillation
* Symptoms of atrial fibrillation
* Referred for catheter ablation

Sub-study:

Same inclusion criteria as the main study plus

-Freedom from arrhythmia the last four days before radiofrequency ablation.

Exclusion Criteria:

* Previous ablation attempts (surgical or catheter ablation)
* Unstable coronary disease
* Heart failure (NYHA III-IV)

Sub-study:

Same exclusion criteria as the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for catheter ablation of atrial fibrillation for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Symptom burden vs. peptide markers for heart failure | 3 years
  Health related quality of life (HRQOL)and arrhythmia symptom burden vill be evaluated and related to the level of four different peptides: NT-pro-BNP, Copeptin, MR-pro-ADM and MR-pro-AMP.
  HRQOL will be measured with the aid of Short-Form-36 (SF-36) and an arrhythmia specific questionnaire containing two parts: One part evaluating symptoms and another part evaluating HRQOL. Both parts are validated and compared to "Symptoms Checklist, Frequency and Severity Scale" and SF-36, respectively.
Sub-study primary outcome: Levels of four biomarkers in relation to heart rhythm | 3 years
  The following biomarkers will be evaluated during sinus rhythm and after at least 30 min of induced atrial fibrillation: NT-pro-BNP, Copeptin, MR-pro-ADM and MR-pro-AMP. These biomarkers will also be measured 24 hours after ablation and at follow-up after three months.

SECONDARY OUTCOMES:
Levels of NT-proBNP and MR-proANP in different sites of the heart and the effect of radiofrequency ablation in relation to heart rhythm | 3 years
  The level of the following biomarkers will be evaluated: NT-pro-BNP, Copeptin, MR-pro-ADM and MR-pro-AMP. These biomarkers will also be measured 24 hours after ablation and at follow-up after three months.
Levels of copeptin and MR-proADM in different sites of the heart and the effect of radiofrequency ablation | 3 years
The relation between left atrial function and neurohormonal activation in patients with atrial fibrillation eligible for radio frequency ablation | 3 years
  The left atrial function is to be echocardiographically accessed. LA volumes , ejection fraction but even 2D strain and strain rate of the left atrium are to be measured. Left ventricular function and left atrial appendix function are also to be studied.
The effect of radiofrequency ablation on the left atrial and left atrial appendix function | 3 years
Alcohol consumption in a atrial fibrillation population undergoing radio frequency ablation (RFA), the connection between alcohol consumption and quality of life and arrhythmia freedom after RFA | 3 years
  Analysis of ethyl glucuronide in hair samples of the patients is to be done in order to access the level of alcohol consumption
Which factors influence the quality of life in patients with atrial fibrillation (AF) undergoing ablation. Do patients with more symptoms have a greater activation of neurohormonal systems and increase of intracardiac pressures after the initiation of AF | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stromberg, Prof, R.N., Principal Investigator — IMH, Dept of Medical and Health Sciences, Linkoping University; Urban Alehagen, Ass prof, MD, Principal Investigator — IMH, Department of Medical and Health Sciences, Linkoping University; Fredrik Nystrom, Prof, M.D., Principal Investigator — IMH, Department of Medical and Health Sciences, Linkoping University; Eva Nylander, Prof, M.D., Principal Investigator — IMH, Department of Medical and Health Sciences, Linkoping University
Locations (1):
- Dept of Cardiology, University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Almroth H, Karlsson LO, Carlhall CJ, Charitakis E. Haemodynamic changes after atrial fibrillation initiation in patients eligible for catheter ablation: a randomized controlled study. Eur Heart J Open. 2023 Oct 31;3(6):oead112. doi: 10.1093/ehjopen/oead112. eCollection 2023 Nov. PMID 38025650
- [Derived] Charitakis E, Karlsson LO, Papageorgiou JM, Walfridsson U, Carlhall CJ. Echocardiographic and Biochemical Factors Predicting Arrhythmia Recurrence After Catheter Ablation of Atrial Fibrillation-An Observational Study. Front Physiol. 2019 Oct 2;10:1215. doi: 10.3389/fphys.2019.01215. eCollection 2019. PMID 31632285
- [Derived] Charitakis E, Barmano N, Walfridsson U, Walfridsson H. Factors Predicting Arrhythmia-Related Symptoms and Health-Related Quality of Life in Patients Referred for Radiofrequency Ablation of Atrial Fibrillation: An Observational Study (the SMURF Study). JACC Clin Electrophysiol. 2017 May;3(5):494-502. doi: 10.1016/j.jacep.2016.12.004. Epub 2017 Mar 1. PMID 29759606
- [Derived] Charitakis E, Walfridsson H, Nylander E, Alehagen U. Neurohormonal Activation After Atrial Fibrillation Initiation in Patients Eligible for Catheter Ablation: A Randomized Controlled Study. J Am Heart Assoc. 2016 Dec 12;5(12):e003957. doi: 10.1161/JAHA.116.003957. PMID 27956398
- [Derived] Charitakis E, Walfridsson H, Alehagen U. Short-Term Influence of Radiofrequency Ablation on NT-proBNP, MR-proANP, Copeptin, and MR-proADM in Patients With Atrial Fibrillation: Data From the Observational SMURF Study. J Am Heart Assoc. 2016 Sep 15;5(9):e003557. doi: 10.1161/JAHA.116.003557. PMID 27633393
- [Derived] Charitakis E, Walfridsson U, Nystrom F, Nylander E, Stromberg A, Alehagen U, Walfridsson H. Symptom burden, Metabolic profile, Ultrasound findings, Rhythm, neurohormonal activation, haemodynamics and health-related quality of life in patients with atrial Fibrillation (SMURF): a protocol for an observational study with a randomised interventional component. BMJ Open. 2015 Dec 21;5(12):e008723. doi: 10.1136/bmjopen-2015-008723. PMID 26692555